CLINICAL TRIAL: NCT04807036
Title: Continuously Iterative Perioperative Holistic Evaluation of Risk and Hypotension Prediction Index
Acronym: CIPHER-HPI
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Edwards Lifesciences (Industry); University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CRI0405
Record Dates: First submitted 2021-03-12; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Surgery--Complications
Keywords: Perioperative medicine; Risk; Predictive analytics; Hypotension Prediction Index; Observational cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Hypotension Prediction Index — HemoSphere Clinical Platform with Acumen Hypotension Prediction Index Feature

SUMMARY:
The investigators would like to explore whether Hypotension Prediction Index during and immediately after surgery can be used to improve the accuracy of scores that predict postoperative problems.

DETAILED DESCRIPTION:
It is known that some patients have a prolonged and difficult recovery after major surgery, which impacts their long-term health and wellbeing. A major issue is that scores for predicting recovery are typically generated only once in the period before surgery, but subsequent events during and immediately after surgery can also alter the likelihood of a prolonged and difficult recovery.

One such event appears to be low blood pressure (hypotension). Hypotension Prediction Index can be calculated from routine blood pressure measurements, and is an indicator of blood pressure instability. The investigators propose that Hypotension Prediction Index during and immediately after surgery may be used to improve their accuracy of scores that predict postoperative problems.

To explore this, the investigators will collect information about the health and care needs, surgery and postoperative recovery of adult patients' requiring major surgery. This data will be taken from hospital information systems, a bedside monitor, test reports, a questionnaire and National Databases. The investigators will then use statistical models to determine whether Hypotension Prediction Index improves the accuracy of preoperative scores for predicting postoperative problems.

Ultimately, the investigators hope to create a tool for predicting how well a patient will recover based on the information available at any given point in time. Healthcare professionals will be able to use this tool to identify and support the needs of patients who need extra help recovering from major surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients who:

1. are referred for CPET
2. are scheduled for elective surgery and expected to have >24 hours postoperative hospital stay
3. will receive invasive arterial pressure monitoring as part of routine care
4. are aged 18 or over
5. have the capacity to give consent to participate

Exclusion Criteria:

Patients who:

1. do not proceed to surgery following CPET referral
2. are aged less than 18 years
3. do not have capacity to consent
4. decline to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are:
  1. referred for routine cardiopulmonary exercise testing
  2. scheduled for elective surgery and expected to have >24 hours postoperative hospital stay
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Days alive and out of hospital | Day 30
  Number of days that the participant is alive and out of hospital

SECONDARY OUTCOMES:
Morbidity | Day 5
  Whether or not a participant has morbidity as measured using the post operative morbidity survey
Complications | From the date and time of surgery until hospital discharge
  Whether or not a participant develops complications as measured using Clavien Dindo
Number of nights that a participant spends at home | Day 30 and 90
Mortality | Day 30 and 1 year
  Number of participants who die within 30 days or 1 year of surgery
Quality of Recovery - 15 score (QoR-15) | Day 90
  A 15 question survey, where a number of different items are scored on a 10 point numeric scale. Higher scores represent better outcomes as reported by the participant
Return to pre-surgery functioning | Day 90
  Participants ability to return to work or usual home activities as measured by item 8 of the Quality of Recovery - 15 score. This will be scored on a 10 point numeric scale. Higher scores represent better outcomes as reported by the patient.
Total length of critical care stay | First 30 days after surgery
  Number of nights spent in Critical Care
Hospital length of stay | Between the date of surgery and hospital discharge (primary admission)
  Number of nights spent in hospital
Hospital readmission | 30 days
  Readmission to hospital following discharge
Total length of hospital stay | 30 days
  Number of nights spent in hospital
Reoperation | Day 30
  Number of unplanned operations

CONTACTS AND LOCATIONS:
Overall Officials: Professor D Levett, Principal Investigator — University Hospital Southampton NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No